CLINICAL TRIAL: NCT03654300
Title: A Volunteer Study to Collect Imaging Data for the Development of the Medaphor Anatomy Guide.
Status: Completed | Type: Observational
Sponsor: Medaphor Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: ML2018_AG_01
Record Dates: First submitted 2018-08-29; First posted 2018-08-31 (Actual); Last update posted 2019-07-25 (Actual); Status verified 2018-08

CONDITIONS: Ultrasound Imaging of Anatomical Structures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of this study is to determine if machine learning can be used to automatically highlight key anatomy on the ultrasound image to help anaesthetists perform ultrasound-guided regional anaesthesia.

DETAILED DESCRIPTION:
The study will involve adult volunteers who are willing to be scanned by a trained sonographer to collect ultrasound video data for the following categories:

* Adductor canal
* Popliteal fossa
* Fascia Iliaca
* Rectus sheath
* Axillary region Each volunteer will be scanned to collect data for every category in the list. Where applicable, both sides of the body will be scanned.

The videos will be segmented by hand to identify the relevant anatomical regions for each category.

The primary objective for this study is to provide the range of data required to develop robust models in conjunction with additional data from patients undergoing a Peripheral Nerve Block procedure that are able to produce the desired segmentation on the unseen validation images. The models will be scored using the standard "Mean intersection over Union" pixel-level metric for semantic segmentation.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, at least 18 years of age;
2. Willing to undergo ultrasound scanning and provide ultrasound video data for the following categories:

   * Adductor canal
   * Popliteal fossa
   * Fascia Iliaca
   * Rectus sheath
   * Axillary region
3. Able to comprehend and sign the Informed Consent prior to enrolment in the study.

Exclusion Criteria:

1. Aged <18 years of age;
2. Unwilling or unable to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers, male and female, aged 18 years or more.
Sampling Method: Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

PRIMARY OUTCOMES:
Model development | 6 months
  models with a Mean intersection over Union score of 0.95 or better for each region in each category.

CONTACTS AND LOCATIONS:
Locations (1):
- Medicentre, Cardiff, United Kingdom